CLINICAL TRIAL: NCT05730907
Title: Efficacy and Clinical Outcomes of Levosimendan in E-CPR
Acronym: ECPR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: MRC-01-21-282
Record Dates: First submitted 2022-12-05; First posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2022-11

CONDITIONS: Cardiogenic Shock; Extracorporeal Membrane Oxygenation Complication
Keywords: levosimendan; ECPR; neurological outcome
MeSH Terms: conditions — Shock, Cardiogenic | interventions — Simendan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Levosimendan — examine whether levosimendan could improve in-hospital survival with good neurological outcomes in patients with cardiac arrest supported by E-CPR

SUMMARY:
Treatment of refractory cardiac arrest requiring cardiopulmonary resuscitation (CPR) may be augmented with Extracorporeal membrane oxygenation (ECMO) to re-establish perfusion in the absence of return of spontaneous circulation. Literature has demonstrated that ECMO initiated during advanced cardiopulmonary life support may confer superior survival rates with acceptable survival and a relatively low incidence of significant neurologic impairment. Levosimendan has not been investigated in patients with cardiac arrest who underwent Extracorporeal CPR (E-CPR). The current study aims to examine whether levosimendan use in the aforementioned patient population could improve survival and ECMO parameters.

ELIGIBILITY:
IInclusion criteria:

* Hospitalized patients ≥ 18 years of age at the time of E-CPR use
* Patients suffered cardiac arrest (IHCA or OHCA)
* Patients received VA-ECMO for E-CPR
* Criteria as per HMC's Extracorporeal Membrane Oxygenation (ECMO) for Cardiac Arrest (E-CPR) clinical practice guidelines (attached with the study protocol)

Exclusion criteria:

* Patients with incomplete key data
* Criteria as per HMC's Extracorporeal Membrane Oxygenation (ECMO) for Cardiac Arrest (E-CPR) clinical practice guidelines (attached with the study protocol)

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study will retrospectively review the electronic medical records of patients who underwent E-CPR at HGH and HH. The units involved are Medical Intensive Care Unit at HGH and both intensive care units at HH i.e., Coronary and Cardiothoracic
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-02-20 (Estimated); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Survival to hospital discharge | 6 months
  Survival to hospital discharge with good neurological outcomes

SECONDARY OUTCOMES:
Survival to decannulation | 6 months
  Survival to decannulation with good neurological outcomes
long term survival | 6 months
  long term survival

CONTACTS AND LOCATIONS:
Overall Officials: Rasha Kaddoura, Principal Investigator — Hamad medical coproation
Locations (1):
- Hamad medical corporation, Doha, DA, Qatar

IPD SHARING:
Plan to Share IPD: No
as per hospital rules and regulations